CLINICAL TRIAL: NCT01071954
Title: An Open Label Study Evaluating the Safety and Efficacy of Long-term Dosing of Romiplostim in Thrombocytopenic Pediatric Subjects With Immune (Idiopathic) Thrombocytopenia Purpura (ITP)
Brief Title: A Study Evaluating the Safety and Efficacy of Long-term Dosing of Romiplostim in Thrombocytopenic Pediatric Patients With Immune (Idiopathic) Thrombocytopenia Purpura
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20090340; 2009-016203-32 (EudraCT Number)
Record Dates: First submitted 2009-12-17; First posted 2010-02-19 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Thrombocytopenia in Pediatric Subjects With Immune Idiopathic Thrombocytopenic Purpura ITP
Keywords: Immune thrombocytopenic Purpura; Pediatric; Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romiplostim (Experimental): Participants received romiplostim administered by subcutaneous injection once a week. The starting dose of romiplostim was 1 μg/kg; weekly dose increases continued in increments of 1 μg/kg/week to a maximum dose of 10 μg/kg in an attempt to reach a target platelet count of between 50 x 10^9/L and 200 x 10^9/L.
  Interventions: Biological: Romiplostim

INTERVENTIONS:
Biological: Romiplostim — Administered by subcutaneous injection once a week.
  Other Names: Nplate

SUMMARY:
This is an extension study designed to assess the safety and durability of platelet count increases with romiplostim treatment of thrombocytopenic patients with immune (Idiopathic) thrombocytopenia purpura. This study is available to pediatric patients who have completed a previous romiplostim ITP study and meet the eligibility criteria of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject or subject's legally acceptable representative has provided informed consent.
* Subject completed a romiplostim study for the treatment of thrombocytopenia in pediatric subjects with ITP.

Exclusion Criteria:

* Subject has or previously had any bone marrow stem cell disorder (any abnormal bone marrow findings other than those typical of ITP must be approved by Amgen before a subject may be enrolled in the study).
* Subject has any new active malignancy diagnosed since enrollment in the previous romiplostim ITP study.
* Subject received any alkylating agents within four weeks before the screening visit or anticipated use during the time of the proposed study.
* Other investigational medications are excluded.
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational agent(s) (with the exception of romiplostim in a previous clinical study).
* Female subject of child bearing potential (defined as having first menses) is not willing to use highly effective contraception during treatment and for 4 weeks after the end of treatment.
* Female subject is pregnant or breast feeding, or planning to become pregnant within 4 weeks after the end of treatment.
* Subject has known sensitivity to any of the products to be administered during dosing.
* Subject previously has entered this study (this will depend on the type of study).
* Subject will not be available for protocol required study visits, to the best of the subject and investigator's knowledge.
* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-12-30 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (29):
- United States (23):
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
- Australia (3):
  - Research Site, Randwick, New South Wales
  - Research Site, South Brisbane, Queensland
  - Research Site, Parkville, Victoria
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Tarantino MD, Bussel JB, Blanchette VS, Beam D, Roy J, Despotovic J, Raj A, Carpenter N, Mehta B, Eisen M. Long-term treatment with romiplostim and treatment-free platelet responses in children with chronic immune thrombocytopenia. Haematologica. 2019 Nov;104(11):2283-2291. doi: 10.3324/haematol.2018.202283. Epub 2019 Mar 7. PMID 30846500
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 28 centers in Australia, Canada, Spain, and the United States. Participants were enrolled from 30 December 2009 until 19 February 2015.
Pre-assignment Details: Pediatric patients who completed a romiplostim study for the treatment of thrombocytopenia in pediatric subjects with immune (idiopathic) thrombocytopenia purpura (ITP) were eligible to participate in this study.
Period: Overall Study
Arm/Group | Romiplostim
Started | 66
Received Treatment | 65
Completed | 39
Not Completed | 27
Not completed — Noncompliance | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 11
Not completed — Requirement for Alternative Therapy | 5
Not completed — Administrative Decision | 5
Not completed — Protocol Specified Criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (4.2)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 37
  Adolescents (12-17 years) | 28
  Adults (18-64 years) | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 29
Race [Count of Participants; unit: Participants]
  White or Caucasian | 40
  Black or African American | 9
  Hispanic or Latino | 9
  Asian | 6
  Japanese | 0
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Aborigine | 0
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The adverse event (AE) severity grading scale used was the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 grading scale, where Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death related to AE.
  A serious adverse event was defined as an adverse event that met at least one of the following serious criteria:
  * fatal
  * life threatening (places the subject at immediate risk of death)
  * required in-patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event. The investigator assessed whether each adverse event was possibly related to the investigational product.
Time Frame: From first dose of study drug until 1 week after last dose. The median (minimum, maximum) duration of treatment was 135.0 weeks (5, 363 weeks).
Population: Enrolled participants who received at least one dose of romiplostim.
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 65
Participants
  All adverse events (AEs) | 64
  Serious adverse events | 19
  AEs leading to discontinuation of study drug | 2
  AEs leading to withdrawal from study | 1
  Grade 3 adverse events | 21
  Grade 4 adverse events | 5
  Grade 5 adverse events | 0
  Treatment-related adverse events (TRAEs) | 17
  Treatment-related serious adverse events | 1
  TRAEs leading to discontinuation of study drug | 0
  TRAEs leading to withdrawal from study | 0
  Grade 3 treatment-related adverse events | 3
  Grade 4 treatment-related adverse events | 1
  Grade 5 treatment-related adverse events | 0

2. Primary Outcome: Duration Adjusted Rate of Treatment Emergent Adverse Events
Description: Exposure adjusted rate was defined as the total number of events divided by the duration of time participants were under observation.
  The adverse event (AE) severity grading scale used was the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 grading scale, where Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death related to AE.
  A serious adverse event was defined as an adverse event that met at least one of the following serious criteria:
  * fatal
  * life threatening (places the subject at immediate risk of death)
  * required in-patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event. The investigator assessed whether each adverse event was possibly related to the study drug.
Time Frame: as for outcome 1
Population: Enrolled participants who received at least one dose of romiplostim.
Measure: Number; unit: events per 100 subject-years
Arm/Group | Romiplostim
Number analyzed (Participants) | 65
events per 100 subject-years
  All adverse events (AEs) | 1397.2
  Serious adverse events | 29.7
  AEs leading to discontinuation of study drug | 2.8
  AEs leading to withdrawal from study | 0.6
  Grade 3 adverse events | 38.5
  Grade 4 adverse events | 6.6
  Grade 5 adverse events | 0.0
  Treatment-related adverse events (TRAEs) | 24.2
  Serious treatment-related adverse events | 1.7
  TRAEs leading to discontinuation of study drug | 0.0
  TRAEs leading to withdrawal from study | 0.0
  Grade 3 treatment-related adverse events | 2.8
  Grade 4 treatment-related adverse events | 0.6
  Grade 5 treatment-related adverse events | 0.0

3. Primary Outcome: Number of Participants Who Developed Antibodies to Romiplostim
Description: Two validated assays were used to test for antibodies to romiplostim / the thrombopoietin-mimetic peptide component of romiplostim (TMP). The first was an immunoassay to confirm the presence of antibodies. The second was a cell-based bioassay to detect neutralizing or inhibitory effects in vitro. If a sample was positive in both assays, a participant was defined as positive for neutralizing antibodies.
  Transient antibodies are those positive post-baseline but negative at the last time point tested.
  Persistent antibodies were those positive at the last time point tested.
Time Frame: Once a year until the end of treatment and 1 week after the end of treatment; median (minimim, maximum) time on study was 34 (2, 91) months.
Population: Enrolled participants who received at least one dose of romiplostim with available postbaseline data
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 64
Participants
  Binding antibodies to romiplostim | 5
  Transient binding antibodies to romiplostim | 4
  Persistent binding antibodies to romiplostim | 1
  Neutralizing antibodies to romiplostim | 1
  Transient neutralizing antibodies to romiplostim | 0
  Persistent neutralizing antibodies to romiplostim | 1

4. Primary Outcome: Number of Participants Who Developed Antibodies to Endogenous Thrombopoietin
Description: Two validated assays were used to test for antibodies to endogenous thrombopoietin (TPO). The first was an immunoassay to confirm the presence of antibodies. The second was a cell-based bioassay to detect neutralizing or inhibitory effects in vitro. If a sample was positive in both assays, a participant was defined as positive for neutralizing antibodies.
  Transient antibodies are those positive post-baseline but negative at the last time point tested.
  Persistent antibodies were those positive at the last time point tested.
Time Frame: as for outcome 3
Population: Enrolled participants who received at least one dose of romiplostim with available postbaseline data
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 64
Participants
  Binding antibodies to TPO | 2
  Transient binding antibodies to TPO | 2
  Persistent binding antibodies to TPO | 0
  Neutralizing antibodies to TPO | 0
  Transient neutralizing antibodies to TPO | 0
  Persistent neutralizing antibodies to TPO | 0

5. Secondary Outcome: Percentage of Participants With a Platelet Response
Description: Platelet response was defined as at least one platelet count ≥ 50 x 10^9/L in the absence of rescue medication during the study.
Time Frame: Assessed every 4 weeks for the duration of treatment; the median (minimum, maximum) duration of treatment was 135.0 weeks (5, 363 weeks).
Population: Enrolled participants who received at least one dose of romiplostim.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 65
percentage of participants | 93.8 (85.0) [85.0 to 98.3]

6. Secondary Outcome: Percentage of Participants Who Used Concomitant ITP Therapy
Time Frame: From baseline to the end of treatment; the median (minimum, maximum) duration of treatment was 135.0 weeks (5, 363 weeks).
Population: Enrolled participants who received at least one dose of romiplostim.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 65
percentage of participants | 47.7 (35.1) [35.1 to 60.5]

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 1 week after last dose. The median (minimum, maximum) duration of treatment was 135.0 weeks (5, 363 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Romiplostim
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 19/65
Other Adverse Events (participants affected / at risk) | 64/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim (N=65)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Mouth haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 3
Ulcer haemorrhage (General disorders) | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Meningitis viral (Infections and infestations) | 1
Metapneumovirus infection (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Haematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim (N=65)
Lymphadenopathy (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Tachycardia (Cardiac disorders) | 4
Ear pain (Ear and labyrinth disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 12
Abdominal pain upper (Gastrointestinal disorders) | 20
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 20
Gingival bleeding (Gastrointestinal disorders) | 13
Gingival pain (Gastrointestinal disorders) | 4
Mouth haemorrhage (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 24
Vomiting (Gastrointestinal disorders) | 32
Chest pain (General disorders) | 4
Fatigue (General disorders) | 15
Injection site bruising (General disorders) | 6
Pain (General disorders) | 8
Pyrexia (General disorders) | 28
Seasonal allergy (Immune system disorders) | 8
Bronchitis (Infections and infestations) | 5
Conjunctivitis (Infections and infestations) | 7
Ear infection (Infections and infestations) | 7
Gastroenteritis viral (Infections and infestations) | 6
Influenza (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 22
Pharyngitis streptococcal (Infections and infestations) | 13
Sinusitis (Infections and infestations) | 5
Tonsillitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 32
Urinary tract infection (Infections and infestations) | 4
Viral infection (Infections and infestations) | 5
Arthropod bite (Injury, poisoning and procedural complications) | 7
Contusion (Injury, poisoning and procedural complications) | 32
Fall (Injury, poisoning and procedural complications) | 5
Head injury (Injury, poisoning and procedural complications) | 5
Laceration (Injury, poisoning and procedural complications) | 10
Ligament sprain (Injury, poisoning and procedural complications) | 7
Limb injury (Injury, poisoning and procedural complications) | 4
Procedural pain (Injury, poisoning and procedural complications) | 6
Scratch (Injury, poisoning and procedural complications) | 7
Skin abrasion (Injury, poisoning and procedural complications) | 15
Decreased appetite (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 11
Joint swelling (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Dizziness (Nervous system disorders) | 11
Headache (Nervous system disorders) | 38
Paraesthesia (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 30
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 31
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 30
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 19
Acne (Skin and subcutaneous tissue disorders) | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 8
Petechiae (Skin and subcutaneous tissue disorders) | 20
Purpura (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 14
Skin lesion (Skin and subcutaneous tissue disorders) | 5
Haematoma (Vascular disorders) | 4
Haemorrhage (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.